CLINICAL TRIAL: NCT03973021
Title: Autologous Very Small Embryonic-like Stem Cells(VSELs) for Organic Erectile Dysfunction
Brief Title: Very Small Embryonic-like Stem Cells for Erectile Dysfunction
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Policy changes have contributed to the failure to carry out smoothly
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Guangzhou Four-Leaf Clover HealthTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VSEL-ED
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-05

CONDITIONS: Organic Erectile Dysfunction
Keywords: erectile dysfunction; very small embryonic-like stem cell
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: In this group, the patients will receive intracavernous injection of autologous VSELs. The check indexes are International Index of Erectile Function 5(IIEF-5), Erection Hardness Score(EHS) and penile vascularization assessed using color duplex Doppler ultrasound (CDDU), mainly including erectile function, stretched penile length, sexual drive, intercourse satisfaction, and overall satisfaction.
Who Masked: Investigator
Masking Description: Different patients receive different numbers of cell for treatment per time
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VSEL Max (Experimental): Each treatment: 120,000 VSELs each time, suspending with 20 mL platelet-rich plasma(PRP), transfusion for 3 times with a interval of 1 month, intracavernous injection
  Interventions: Biological: Very small embryonic-like stem cell(VSEL)
- VSEL Medium (Experimental): Each treatment: 90,000 VSELs each time, suspending with 20 mL platelet-rich plasma(PRP), transfusion for 3 times with a interval of 1 month, intracavernous injection
  Interventions: Biological: Very small embryonic-like stem cell(VSEL)
- VSEL Mini (Experimental): Each treatment: 60,000 VSELs each time, suspending with 20 mL platelet-rich plasma(PRP), transfusion for 3 times with a interval of 1 month, intracavernous injection
  Interventions: Biological: Very small embryonic-like stem cell(VSEL)
- Control (No Intervention): In this group, the patients will receive 20 mL platelet-rich plasma(PRP) treatment and as a control group.

INTERVENTIONS:
Biological: Very small embryonic-like stem cell(VSEL) — Mononuclear cells were collected from peripheral blood of each patient using a machine, VSELs were isolated, and each group was injected according to different numbers after activation
  Arms: VSEL Max; VSEL Medium; VSEL Mini

SUMMARY:
The aim of this study is the safety and efficacy of autologous very small embryonic-like stem cells(VSELs) to organic erectile dysfunction, such as those associated with metabolic syndrome or the treatment of prostate cancer.

DETAILED DESCRIPTION:
By enrolling patients with organic erectile dysfunction adapted to enrolled criteria, this study will document for the first time the safety and efficacy of underlying penile cellular damage.

The safety will be evaluated by tolerance degree. The efficacy will be evaluated validated scores and color duplex Doppler ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic and systemic changes in diseases such as diabetes and atherosclerosis or more localized causes such as direct injury to the penile neurovascular supply during prostate surgery
* Diagnosed as an organic erectile dysfunction by at least 2 urological surgeons

Exclusion Criteria:

* Non-organic erectile dysfunction, such as psychological factors
* Solid cancer patients other than early prostate cancer
* Blood disease patients, thrombocytopenia or dysfunction, hypofibrinogenemia or anticoagulant therapy, long-term use of aspirin
* Older than 70 years

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Tolerance | 1-4 weeks after each injection
  Evaluation indicators include postoperative pain at the injection site (VAS score), hematoma, abscess, or priapism

SECONDARY OUTCOMES:
Short-term effects on erectile function | 3-6 months after each injection
  Assessment using International Index of Erectile Function 5, which is physicians global assessment to measure erectile function
Long-term effects on erectile function | 12 months after final injection
  Assessment using International Index of Erectile Function 5, which is physicians global assessment to measure erectile function

CONTACTS AND LOCATIONS:
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No